CLINICAL TRIAL: NCT03914690
Title: Effect of Erythropoietin on Neurodevelopmental Outcomes in Very Preterm Infants With Intraventricular Hemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhengzhou University (Other)
Collaborators: Zhengzhou Children's Hospital, China (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Changlian Zhu, Director, Clinical research center, Third Affiliated Hospital of Zhengzhou University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EPO2014
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Premature Infants
MeSH Terms: conditions — Premature Birth | interventions — Erythropoietin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythropoietin (Experimental): EPO is administered 500IU/kg, intravenously after diagnosis of IVH within 72h after birth, and every other day for 2 weeks. Recombinant human erythropoietin was configured by the hospital pharmacy intravenous Centre Configuration, melted configured with saline to 1ml/kg solution.
  Interventions: Drug: Erythropoietin
- Normal saline (Placebo Comparator): Normal saline is administered the same volume with EPO, intravenously after diagnosis of IVH within 72h after birth, and every other day for 2 weeks.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Erythropoietin — EPO is administered 500IU/kg, intravenously after diagnosis of IVH within 72h after birth, and every other day for 2 weeks.
  Other Names: Epoietin Beta
  Arms: Erythropoietin
Drug: Normal saline — Normal saline is administered the same volume with EPO, intravenously after diagnosis of IVH within 72h after birth, and every other day for 2 weeks.
  Arms: Normal saline

SUMMARY:
Erythropoietin (EPO) has been shown to be neurotrophic and neuroprotective in several animal models and some clinical studies. Our hypothesis is that EPO could improve long-term neurological outcomes in very preterm infants with intraventricular hemorrhage (IVH). The aim of this study is to evaluate the long-term neuroprotective effect of repeated low-dose EPO (500 U/kg) in very preterm infants with IVH.

DETAILED DESCRIPTION:
IVH is one of the most common complications in preterm infants. Nearly 60% of preterm infants with grade III-IV IVH develop severe neurodevelopmental outcomes. There are currently no effective treatments to prevent preterm infants with IVH from developing ventricular dilation or serious neurological disabilities. Recent studies have shown that EPO could improve neurodevelopmental outcomes in preterm infants with grade III-IV IVH. However, the dose and course of EPO in preterm infants is still uncertain. The purpose of the study was whether repeated low-dose EPO (500 U/kg, every other day, for 2 weeks) given to very preterm right after the diagnosis of IVH could improve long-term neurological outcomes. Very preterm infants with gestational age of ≤ 32 weeks who are diagnosed with IVH within 72 hours after birth in NICU are eligible for enrolment. After informed consent is obtained, infants will be randomly assigned to EPO group or vehicle group. The primary outcome is whether EPO improves mortality and neurological disabilities in very preterm infants with IVH at 18 months of corrected age, and the secondary outcome was whether EPO decrease the incidence of cerebral palsy, MDI<70, blindness, and deafness.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants admitted to NICU ≤ 32 weeks gestation at birth
* Birth weight less than 1500 g
* Less than 72 hours of life at time of enrolment
* Diagnosed as IVH by head ultrasound
* Written informed consent of parent or guardian

Exclusion Criteria:

* Genetic metabolic diseases
* Congenital abnormalities
* Polycythaemia (Hct > 65%) within first 24 hours of life
* Thrombocytopenia (platelets < 50K cells/microL) within first 24 hours of life
* Unstable vital signs (such as respiration and circulation failure)

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Mortality | At corrected age of 18 months
  To compare the death rate in EPO treatment and control groups at 18 months of corrected age.
Incidence of neurological disability | At corrected age of 18 months
  To evaluate neurodevelopmental function via Bayley Infant Development scale (2nd Edition), visual acuity and auditory brainstem response measurements at 18 months of corrected age.

SECONDARY OUTCOMES:
Incidence of cerebral palsy | At corrected age of 18 months
  To compare the incidence of cerebral palsy in EPO treatment and control groups at 18 months of corrected age.
Incidence of MDI<70 | At corrected age of 18 months
  To compare the incidence of MDI<70 via Bayley Infant Development scale (2nd Edition) in EPO treatment and control groups at 18 months of corrected age.
Incidence of blindness | At corrected age of 18 months
  To compare the incidence of blindness via visual acuity and sight radius examinations in EPO treatment and control groups at 18 months of corrected age.
Incidence of deafness | At corrected age of 18 months
  To compare the incidence of deafness via auditory brainstem response measurements in EPO treatment and control groups at 18 months of corrected age.
The effect of EPO treatment on blood mRNA expression | At 3 weeks after birth
  To investigate different mRNA expression between EPO and control group, peripheral venous blood of preterm infants after EPO treatment will be collected in both EPO group and control group, and the transcriptome of the premature infant blood will be assayed by RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Changlian Zhu, PhD, Study Chair — Third Affiliated Hospital of Zhengzhou University
Locations (1):
- Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song J, Wang Y, Xu F, Sun H, Zhang X, Xia L, Zhang S, Li K, Peng X, Li B, Zhang Y, Kang W, Wang X, Zhu C. Erythropoietin Improves Poor Outcomes in Preterm Infants with Intraventricular Hemorrhage. CNS Drugs. 2021 Jun;35(6):681-690. doi: 10.1007/s40263-021-00817-w. Epub 2021 May 6. PMID 33959935